CLINICAL TRIAL: NCT02021448
Title: Predictive Factors of Obesity-hypoventilation Syndrome (OHS) Among Obese Subjects- ETUDE COHYPOB -
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty in recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5059
Record Dates: First submitted 2013-08-29; First posted 2013-12-27 (Estimated); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Obesity-hypoventilation Syndrome; Nocturnal Alveolar Hypoventilation
Keywords: OHS
MeSH Terms: conditions — Obesity Hypoventilation Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Obesity: BMI > 30 kg/m2 (Other): Annual visits among 3 years. During each visit different testings are performed in order to detect an obesity-hypoventilation syndrome (OHS) Polygraphy/Polysomnography, Blood sampling, EKG, Lung function testing, Arterial blood gases, Thoracic radiography, Six-minute walk test, Respiratory questionnaires
  Interventions: Other: Annual visits among 3 years. During each visit different testings are performed in order to detect an obesity-hypoventilation syndrome (OHS)

INTERVENTIONS:
Other: Annual visits among 3 years. During each visit different testings are performed in order to detect an obesity-hypoventilation syndrome (OHS) — Polygraphy/Polysomnography,Blood sampling, EKG,Lung function testing,Arterial blood gases,Thoracic radiography,Six-minute walk test,Respiratory questionnaires

SUMMARY:
Investigate whether the course of an isolated nocturnal alveolar hypoventilation can predict the future occurrence of obesity-hypoventilation syndrome (OHS) in obese subjects

ELIGIBILITY:
Inclusion criteria:

* Obese volunteer Subject (BMI> 30 kg/m2)
* Adults of either sex
* Social security affiliation
* Written informed consent

Exclusion criteria:

* Confirmed OHS at baseline defined by a daytime hypercapnia with PaCO2> 45mmHg
* Any cause of chronic respiratory failure other than obesity such as COPD, chest deformation, phrenic nerve paralysis, pulmonary fibrosis, neuromuscular disease, a history of mutilating thoracic surgery ...
* Obstructive ventilatory defect with FEV1/ FVC <70% post-bronchodilator
* Long term oxygen therapy, noninvasive ventilation, continuous positive airway pressure
* Any serious illness involving life-threatening within 3 years after inclusion
* Drug or alcohol abuse
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2022-01 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Occurrence of obesity-hypoventilation syndrome | 3 years
  partial pressure of carbon dioxide in the arterial blood > 45mmHg

CONTACTS AND LOCATIONS:
Overall Officials: KESSLER Romain, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (6):
- France (6):
  - CHU Angers, Angers
  - CHU Brest, Brest
  - CH Cannes, Cannes
  - CHU Grenoble, Grenoble
  - CHU Reims, Reims
  - CHU Strasbourg, Strasbourg